CLINICAL TRIAL: NCT05026047
Title: Acceptability of Human Papillomavirus Self-sampling in Women Living With HIV
Acronym: AUTOCol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: APHP200078
Record Dates: First submitted 2021-04-29; First posted 2021-08-30 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Papillomavirus Infection
Keywords: Smear test; Early detection of cancer; Papillomavirus infection; Vaginal self-sampling
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients consulting in an infectious disease department (Experimental): no comparator
  Interventions: Other: HPV self-sampling

INTERVENTIONS:
Other: HPV self-sampling — HPV self-sampling in HIV-positive women

SUMMARY:
Women living with HIV are unsufficiently screened for cervix cancer although they have a higher risk of developping it, resulting in many obstacles. Offering a new screening technique, more accessible and which doesn't require gynecologic examination, could help improving this coverage rate. Human Papillomavirus (HPV) screening have a higher-performance for cervix cancer than smear test. Self-collected vaginal swabs are as efficient as vaginal swabs performed by clinicians. They are also shown as acceptable among general population but only one study in South Africa has been performed on women living with HIV. In addition, recent studies on urine self-sampling for high risk HPV (HR-HPV) screening report satisfactory performance. The main hypothesis is that self-collected vaginal swabs and urine self-sampling are also acceptable among women living with HIV in the CoreVIH Ile de France Nord (CoreVIH) cohort.

DETAILED DESCRIPTION:
Worldwide, cervical cancer is the second most common cancer (10% of all cancers), in 2012: 528,000 cases and 266,000 deaths. In France, in 2012, the incidence is estimated at 6.7 per 100,000 women, with 3,028 new cases per year and 1,102 deaths. Screening for cervical cancer is a public health issue because cancer affects young, healthy women and early detection is available. Persistent infection with oncogenic HPV (Human Papillomavirus) is responsible for the development of pre-cancerous lesions and cervical cancer. There are more than a hundred genotypes of HPV identified. Among them, HPV 16 and 18 are the genotypes most often associated with cancer. The natural history of cervical cancer has led to the definition of several ways to prevent the development of cancer, such as vaccination to prevent infection, screening for infection using HPV virological tests that detect DNA, and cervical smears to detect precancerous or cancerous lesions. In France, in the general population, screening is done by smear test performed by a clinician or in a biological laboratory for cytological analysis. The recommendations of the French Health Authority (HAS) are to perform a smear test every three years, after two normal smears one year apart from 25 to 65 years of age, except in women who have never had sexual intercourse and those who have had a hysterectomy with removal of the cervix. Since July 2019, the HAS has introduced in its recommendations for cervical cancer screening the use of HPV testing, which must now replace the cytological examination from the age of 30 years and must be performed 3 years after the last cytological examination with a normal result and then every 5 years in case of negativity.

This test can be offered as a vaginal self-sampling for women who are not or insufficiently screened. Women living with HIV are part of this population and are included in these recommendations. Other countries such as the Netherlands have included virological analysis in their strategy: in 2011 the health authorities have decided to use HPV self-tests in primary care instead of cervical smear tests (FCU). In 2016, the recommendation in the Netherlands is to perform an HPV test every 5 years from 30 to 60 years of age. In case of a positive HPV test, an FCU is performed.

Virological tests can be carried out on vaginal swabs by hetero or self-sampling or on urine samples. In HIV patients, earlier screening is recommended because of the increased risk of developing cancerous lesions as a result of immunosuppression. The Morlat report (2013) recommends an annual smear test as soon as seropositivity is discovered, with no upper age limit. France has individual and unorganized screening (such as breast or colon cancer) with incomplete coverage. According to HAS data in 2010, only 8% of women eligible for smear screening have an adequate follow-up rate. 52% of women aged 25-65 are not screened at all or have smears too far apart (more than 3 years). A majority of cases of cervical cancer are diagnosed in France in women participating irregularly or not participating in individual screening. The tests are based on the detection of HPV on a sample of the cervix. The virological technique is already recommended in the triage of smear test with atypical squamous cells of undetermined significance (ASC-US). Several types of self-samples are currently available. Studies show a good level of agreement for all vaginal swabs using HPV testing by polymerase chain reaction (PCR) technique (dry swab, swab with liquid transport medium). The different studies that have tested the acceptability of HPV self-sampling in the general population show good acceptability; between 66 and 94% acceptability depending on the studies.

The use could be interesting in the first instance to catch up with women who have not been screened due to the hindrance of gynaecological examination or the constraint of a medical consultation. In a French study, the APACHE project, the proposal of self-sampling in unscreened women had increased participation in cervical cancer screening. The use of self-sampling improves participation in screening by sending the kits to women who are not up-to-date in their smear test. In a study conducted among HIV-infected women in South Africa in 2015, there was 90% acceptability.

The APACHE project is a series of studies carried out in France between 2009 and 2014 on the subject whose two objectives were to evaluate the performance of self-sampling for the detection of cervical HPV infection and to assess the effectiveness on participation of sending a self-sampling kit to the homes of undetected women.

A previous medical thesis showed that 54% of patients followed up at the CoreVIH Ile de France Nord had a smear that was less than two years old (9). The idea is therefore to explore alternative options for these women who are being followed at CoreVIH Ile de France Nord but who are not being screened at the recommended rate.

ELIGIBILITY:
Inclusion criteria :

* HIV-positive women over or equal to 30 years old
* HIV-positive patient who has already consulted at least once at the CoreVIH Ile de France Nord

Exclusion criteria :

* Refusal to sign a consent form
* Personal history of cervical cancer, conization, suspicious smears undergoing exploration or known high oncogen risk HPV
* Ongoing menstruation
* Physical impossibility to carry out self-sampling (e.g. motor disability, significant visual disturbances)
* Ongoing gynecological infection
* Patient not affiliated to a social security scheme or without AME
* Protected adult patient (under guardianship, curatorship)
* Pregnant or breastfeeding woman

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — HIV-positive women
Enrollment: 200 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Acceptability of vaginal self-test coupled to urinary self-sampling in HIV-positive women in the population of the CoreVIH Ile de France Nord area. | one day
  Percentage of refusals to perform both tests.

SECONDARY OUTCOMES:
Acceptability of the vaginal self-test alone and the urinary self-sampling alone in HIV-positive women in the population of the CoreVIH Ile de France Nord area. | one day
  Percentage of refusal to perform vaginal or urinary self-sampling
Evaluation of the quality of vaginal self-test | one day
  Quantification of cellularity in vaginal self-tests
Prevalence of HR-HPV in both samples (vaginal self-test and/or urinary self-sampling) | one day
  Number of tests positive to at least one HPV-HR compared to the number of tests performed and interpretable
Factors associated with the acceptability of self-sampling (vaginal self-test and/or urinary self-sampling) | one day
  The acceptability of the self-sampling will be evaluated by the participants' answers to a standardized questionnaire (anxiety about finding abnormal results, preference for sample collection by a physician, fear of injury). The individual factors suspected of being associated with acceptability will be compared between the two groups.
Feasibility in carrying out self-sampling | one day
  The feasibility of self-sampling will be evaluated by the participants' answers to a standardized questionnaire on their feelings during the self-sampling: sensation at the time of the test, comfort and pain.

CONTACTS AND LOCATIONS:
Overall Officials: Morgane MAILHE, MD, Principal Investigator — AP-HP SMIT, Bichat hospital, Paris, France
Locations (1):
- Hôpital Bichat, SMIT, Paris, Île-de-France Region, France